CLINICAL TRIAL: NCT07009262
Title: A Prospective, Non-interventional Study in Patients With Type I or II Hereditary Angioedema Using Icatibant for On-demand Treatment of Attacks
Brief Title: A Study Observing US Patients With HAE Type I or II Who Take Icatibant to Treat HAE Attacks
Acronym: ICTOS
Status: Completed | Type: Observational
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Collaborators: US Hereditary Angioedema Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: ICTOS-001
Record Dates: First submitted 2025-05-07; First posted 2025-06-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with Type I or II Hereditary Angioedema Using Icatibant for On-demand Treatment of Attacks.
  Interventions: Other: Inapplicable

INTERVENTIONS:
Other: Inapplicable — Inapplicable

SUMMARY:
Patients with HAE Type I or II who enroll in the study are asked to complete a patient diary when they experience an HAE attack. If icatibant is taken as the first treatment for the attack, the patient diary will ask questions over a 48 hour period after dosing to track the characteristics and severity of the attack along with the patient's level of anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 12 years of age and older
2. Diagnosis of HAE Type I or II, based on US Hereditary Angioedema Association (HAEA) database records and/or verbal confirmation from the patient
3. Currently using icatibant to treat HAE attacks
4. If a patient is receiving long-term prophylactic treatment, they must have been on a stable dose and regimen for at least 3 months prior to the Screening Visit
5. Patient has had at least 2 HAE attacks in the 3 months prior to the Screening Visit, as self-reported verbally by the patient
6. Patient is able to read, understand, and complete the eDiary
7. Patient is willing and able to adhere to all protocol requirements

Exclusion Criteria:

1. Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1-inhibitor deficiency, HAE with normal C1-INH (previously known as HAE Type III), idiopathic angioedema, or angioedema associated with urticaria
2. Use of angiotensin-converting enzyme inhibitors
3. Participation in any gene therapy treatment or trial for HAE
4. Participation in any interventional investigational clinical trial within 4 weeks prior to screening
5. Any pregnant or breastfeeding patient

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a self-reported diagnosis of HAE Type I or II who take icatibant to treat HAE attacks
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGI-C) | Within 12 hours of the first Icatibant dose adminstration
  time to beginning of symptom relief defined as at least ''a little better'' (2 time points in a row)

SECONDARY OUTCOMES:
Patient Global Impression of Severity (PGI-S) | Within 12 hours of the first Icatibant dose adminstration
  Time to first incidence of decrease from baseline (2 time points in a row)
PGI-S: Time to Complete HAE Attack Resolution | Within 24 hours of the first Icatibant dose adminstration
  time to HAE attack resolution, defined as ''none''
Return to normal function | At 48 hours after first Icatibant dose adminstration
  Time to return to normal daily activities. Date/Time or one of the following options:
  * Not Applicable - daily activities were not affected
  * not yet returned to normal activities
General Anxiety Numeric Rating Scale (GA-NRS): Cumulative GA-NRS | over 12 and 24 hours of the first icatibant administration
  Patient is asked 'How anxious do you feel right now?' 11-point numeric scale, 0-10 with 0=Not at all anxious and 10=Extremely anxious

CONTACTS AND LOCATIONS:
Locations (1):
- KalVista Investigative Site, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing but only after deidentification of individual patient data.